CLINICAL TRIAL: NCT01310504
Title: The Use of the FAST Scan by Paramedics in Mass Casualty Incidents
Brief Title: The Use of the FAST (Focused Abdominal Scan for Trauma) Scan by Paramedics in Mass Casualty Incidents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, J. Andrew Cusser, MD, Ascension Health
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ME 10 0050
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Mass Casualty

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non peritoneal dialysis patient (Active Comparator)
  Interventions: Procedure: SonoSite Ultrasound
- Peritoneal dialysis patient (Active Comparator)
  Interventions: Procedure: SonoSite Ultrasound

INTERVENTIONS:
Procedure: SonoSite Ultrasound — Will be moulaged to resemble a peritoneal dialysis patient. Paramedics will scan the abdomen and determine it there's fluid within.
  Arms: Non peritoneal dialysis patient
Procedure: SonoSite Ultrasound — Paramedics will scan the abdomen and determine it there's fluid within.
  Arms: Peritoneal dialysis patient

SUMMARY:
Initially a group of paramedics will be trained to perform FAST (Focused Abdominal Scan for Trauma) scans. The paramedics will then enter a simulated mass causality incident and triage patients. Volunteers in the study will include peritoneal dialysis patients ("non stable") and non-peritoneal dialysis patients ("stable"). They will use the ultrasound to perform FAST scans on the patients to determine which subjects are "stable" and which are "unstable" patients. They will record which patients they consider need transport first. This data will be used to evaluate accuracy and speed of the FAST scan. When the paramedic identifies free fluid within the volunteer, they will be able to make the decision to upgrade these patients and ultimately transport them more quickly. The paramedics will be evaluated for time and accuracy with the FAST scan.

DETAILED DESCRIPTION:
Ultrasound and the FAST (Focused Abdominal Scan for Trauma) scan is currently being used in the Emergency Department to help evaluate trauma patients. In the field a paramedic will use the START (Simple Triage Rapid Treatment) triage procedure to evaluate many patients and to help decide which patients are more critical and therefore need to be transported first. This study aims to create a mass casualty environment through the use of 10 volunteers who are on peritoneal dialysis and 10 patients who are not.

ELIGIBILITY:
Inclusion Criteria:

Paramedic - at least one year in the field, physically able to perform the test

Patients:

* (10)peritoneal dialysis patient that are able to leave dialysate in abdominal cavity for the duration of the test
* (10) subjects not on peritoneal dialysis who are available for the duration of the test

Exclusion Criteria:

* Under 18 years of age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the use of the ultra sound and FAST scans in a simulation of a mass causality incident by paramedics for accuracy and speed | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: James A Cusser, MD, Principal Investigator — Ascension Health
Locations (1):
- Genesys Regional Medical Center, Grand Blanc, Michigan, United States